CLINICAL TRIAL: NCT02238678
Title: Impact of Deep Endometriosis Surgery on Bladder Function
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Department of Obstetrics and Gynaecology, Insubria Unievrsity, Varese (Italy) (Unknown)
Responsible Party: Principal Investigator, Laterza Rosa Maria, Dr. med, Medical University of Vienna
Other Study IDs: ENDOBLAD 1057/2014
Record Dates: First submitted 2014-08-28; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-08

CONDITIONS: Deep Infiltrating Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Deep endometriosis patients

SUMMARY:
It has been demonstrated that ligaments, both cardinal and uterosacral contain a considerable amount of autonomic nerve tissues. The resection of deep infiltrating endometriotic nodules at the level of the uterosacral ligaments or the rectovaginal space is supposed to damage the supplying autonomic nerve fibers of the lower urinary tract. The bladder receives motor and sensitive innervations from both the sympathetic fibers, most of which arise from the hypogastric plexuses and nerves, and the parasympathetic fibers, which arise from the pelvic splanchnic nerves and the inferior hypogastric plexus; therefore, even bladder function may be impaired in women affected by deep endometriosis.

Very few data have been published regarding the urodynamic functional evaluation of bladder in patient with deep endometriosis.So far, it is unknown if the surgery itself causes the postoperative bladder dysfunction or if the surgery unmasks a subclinically pre-existing detrusor pathology.

Since the urinary postoperative complications have a strong impact on quality of life of the deep endometriosis patients and often requires management (due to a poor spontaneous remission), it is crucial a better understanding of the problem. That will help for a more appropriate pre-operative counselling.

Aims of this study are to evaluate the bladder function before and after deep endometriosis surgery, using standardized validated instruments and to correlate the localisation of the endometriosis lesion, the type/area of surgical dissection with the postoperative bladder function.

This is a prospective multicenter cohort study involving the Department of General Gynaecology and Gynecological Oncology of Medical University of Vienna (Austria) and the Department of Obstetrics and Gynaecology of Insubria University, Varese (Italy).

A total of 50 patients are planned to be included. The study protocol consider a Preoperative Assessment (clinical examination, transvaginal pelvic ultrasound, preoperative specific questionnaire including obstetric, medical, and surgical history and standardized questions on pelvic floor dysfunctions, standardized instrumental assessment of the pelvic floor) a Intraoperative Assessment (during laparoscopy, the localizations of endometriotic lesions recorded and identified by anatomical sites, numbers, and depth of infiltration). Before and 3 months after surgery a Urodynamic assessment is planned.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of deep infiltrating endometriosis requiring surgical treatment
* Patient planned to be submitted to laparoscopic surgery finalize to eradicate the endometriosis pathology
* Naïve patients for OAB treatment.
* Patients must be capable of independent toileting
* Patients must be able to fully understand all study procedures and to provide written informed consent to study participation

Exclusion Criteria:

* Patient previously submitted to pelvic surgery for any urogynaecological disease;
* Patients previously submitted to DE surgery
* Patient with documented clinical, instrumental, or laparoscopic preoperative diagnosis of bladder endometriosis;
* Patient with documented urinary tract infection
* Patient with history of diabetes mellitus, psychiatric, or neurological disease;
* Pregnant patients
* Patients < 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients with confirmed diagnosis of deep infiltrating endometriosis requiring surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Urodynamic assessment after deep infiltrating endometriosis surgery | 2 years
  to evaluate the bladder function before and after deep endometriosis surgery (Unit of Measure: First Desire (ml) from Urodynamic Assessment)

SECONDARY OUTCOMES:
Bladder symptoms after surgery for deep infiltrating endometriosis | 2 years
  using standardized validated questionnaires -OABQ short form, ICIQ short form questionnaire, micturition diary.
correlation between localisation of the endometriosis lesion and postoperative bladder function. | 2 years
  to correlate the localisation of the endometriosis lesion, the type/area of surgical dissection with a specific urodynamic pattern and/or a specific low urinary tract symptom

REFERENCES:
- [Derived] Laterza RM, Uccella S, Serati M, Umek W, Wenzl R, Graf A, Ghezzi F. Is the Deep Endometriosis or the Surgery the Cause of Postoperative Bladder Dysfunction? J Minim Invasive Gynecol. 2022 Apr;29(4):567-575. doi: 10.1016/j.jmig.2021.12.017. Epub 2022 Jan 2. PMID 34986409